CLINICAL TRIAL: NCT04046341
Title: Implementing Evidence-based Behavioral Sleep Intervention in Urban Primary Care: Aim 2
Brief Title: Implementing Behavioral Sleep Intervention in Urban Primary Care
Acronym: Aim_2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-016482
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Results first posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Sleep Disturbance; Sleep Deprivation; Sleep
Keywords: Difficulty falling asleep; Difficulty staying asleep; Not getting enough sleep
MeSH Terms: conditions — Parasomnias; Sleep Deprivation

STUDY DESIGN:
Intervention Model Description: Caregiver-child dyads (child ages 1-5 years with a sleep problem) will be recruited from CHOP urban primary care sites.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Sleep Intervention (Experimental): Parents attend 1-3 one-hour sessions at their primary care office or via telemedicine, where they receive sleep education and work with interventionists to develop strategies to help their child at bedtime.
  Interventions: Behavioral: Sleep Well!

INTERVENTIONS:
Behavioral: Sleep Well! — The intervention comprehensively addresses poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers. Interventionists will use strategies to engage with and empower families, such as motivational interviewing and collaborative problem-solving. Session content will be reinforced via phone calls from interventionists. Families will receive intervention session appointment reminders and information about intervention content (e.g., reminders to follow a bedtime routine) via text message.

SUMMARY:
Investigators will enroll up to 20 participants from 3 Children's Hospital of Philadelphia (CHOP) primary care locations. The primary objective is to determine the whether the Sleep Well! behavioral sleep intervention is feasible to be implemented in primary care offices and acceptable to families. The direction and magnitude of change in child sleep from pre-intervention to post-intervention will also be examined.

DETAILED DESCRIPTION:
Behavioral sleep problems such as insomnia and insufficient sleep are common in toddlers and preschoolers and disproportionately impact lower socioeconomic status (SES) children. Despite a robust evidence base, behavioral sleep interventions are rarely tested with lower-SES children or in primary care, an accessible service delivery setting. The primary objective of this study is to determine the whether the Sleep Well! behavioral sleep intervention is feasible and acceptable to families. We will also examine the direction and magnitude of change in child sleep from pre-intervention to post-intervention. This is a preliminary open trial of the Sleep Well! program with pre-intervention and post-intervention assessments.Caregiver-child dyads (child ages 1-5 years with a sleep problem) will be recruited from CHOP urban primary care sites.

Sleep Well! is a brief, behavioral sleep intervention for toddlers and preschoolers who have a caregiver-reported sleep problem or who are not getting enough sleep. The intervention includes evidence-based behavioral sleep approaches and strategies to engage and empower families. The primary outcomes for this open trial are feasibility (number of caregivers recruited, engaged, and retained in intervention; participant intervention attendance rate) and caregiver acceptability, assessed via a questionnaire and qualitative post-intervention interview. Secondary outcomes are the direction and magnitude in any pre- to post-intervention change in child sleep.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver participant is the parent or legal guardian of the child subject.
* Caregiver/legal guardian 18 years of age.
* Child between the ages of 1 and 5 years.
* Presence of caregiver-reported child sleep problem determined by a Brief Child Sleep Questionnaire item, included in an eligibility screening questionnaire or child meets American Academy of Sleep Medicine diagnostic criteria for either pediatric insomnia or insufficient sleep, assessed through an eligibility screening questionnaire.
* English-speaking.

Exclusion Criteria:

* Caregiver is not parent or legal guardian of child participant.
* Presence of a diagnosed child neurodevelopmental (e.g., autism spectrum disorder; Trisomy 21) or chronic medical condition (e.g., sickle cell disease, cancer) in which the disorder or treatment of the disorder impact sleep.
* Caregivers/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Williamson, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williamson AA, Okoroji C, Cicalese O, Evans BC, Ayala A, Harvey B, Honore R, Kratchman A, Beidas RS, Fiks AG, Power TJ, Mindell JA. Sleep Well! An adapted behavioral sleep intervention implemented in urban primary care. J Clin Sleep Med. 2022 Apr 1;18(4):1153-1166. doi: 10.5664/jcsm.9822. PMID 34910624

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Both caregivers and children were enrolled in the study and were combined as a dyad.
Groups:
- Behavioral Sleep Intervention: Caregivers attend 1-3 one-hour sessions at their primary care office or via telemedicine, where they receive sleep education and work with interventionists to develop strategies to help their child at bedtime.
  Sleep Well!: The intervention comprehensively addresses poor sleep health behaviors (e.g., use of electronics at bedtime; inconsistent and variable sleep schedules; lack of a bedtime routine) as well as insomnia (difficulty falling and staying asleep; the need for caregiver presence at bedtime) and insufficient sleep in toddlers and preschoolers. Interventionists will use strategies to engage with and empower families, such as motivational interviewing and collaborative problem-solving. Session content will be reinforced via phone calls from interventionists. Families will receive intervention session appointment reminders and information about intervention content (e.g., reminders to follow a bedtime routine) via text message.
Period: Overall Study
Arm/Group | Behavioral Sleep Intervention
Started | 15
Completed | 12
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: At baseline, we collected data from 15 caregiver-child dyads that initiated the intervention. Three families were lost to follow-up so post-intervention data were collected from 12 caregiver-child dyads.
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants] — Categorical age is presenting for caregiver participants in the caregiver-child dyads who participated.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 15
    >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Continuous age information is based on the child participant in the caregiver-child dyad.
  years | 3.00 (1.36)
Sex: Female, Male [Count of Participants; unit: Participants] — This information is for the child participants in the caregiver-child dyad.
  Participants
    Female | 11
    Male | 4
Sex: Female, Male [Count of Participants; unit: Participants] — This information is for the caregiver participant in the caregiver-child dyad.
  Participants
    Female | 15
    Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This information is for the child in the caregiver-child dyad.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 14
    Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This information is for the caregiver in the caregiver-child dyad
  Participants
    Hispanic or Latino | 2
    Not Hispanic or Latino | 13
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — This information is for the child in the caregiver-child dyad.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 13
    White | 2
    More than one race | 0
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — This information is for the caregiver in the caregiver-child dyad
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 12
    White | 2
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
Brief Child Sleep Questionnaire- Perceived Sleep Problem [Count of Participants; unit: Participants] — Questionnaire item for Brief Child Sleep Questionnaire that asks caregivers about the severity of a child sleep problem. A very small or no sleep problem is coded as 0, and a small to severe sleep problem is coded as 1.
  Participants
    Caregiver-perceived sleep problem | 15
    No caregiver-perceived sleep problem | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Caregiver-child Participants Who Complete All Intervention Procedures Following Enrollment (Retention Rate)
Description: The study team will track the number of caregiver-child dyad participants who complete all intervention procedures following enrollment.
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 15
Participants
  Retained in intervention | 13
  Attrition from intervention | 2

2. Primary Outcome: Number of Caregiver-child Participants Who Complete All Assessments (Pre-intervention and Post-intervention) That Were Planned (Feasibility)
Description: The study team will track the number of proportion of participants who complete all assessments (pre-intervention and post-intervention) that were planned.
Time Frame: Approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 15
Participants
  All assessments completed | 12
  Post-intervention assessment not completed | 3

3. Primary Outcome: Treatment Acceptability (Strategies)
Description: Caregivers will complete the Treatment Evaluation Inventory-Short Form, a widely used measure of treatment acceptability that has been adapted for the purposes of the Sleep Well! intervention. Ratings are shown for proportion of caregivers agreeing or strongly agreeing with the statement that the strategies are acceptable.
Time Frame: 3 months
Population: The treatment evaluation form was administered at post-intervention only and thus data were not available for the 3 participants who did not complete the post-intervention assessment.
Measure: Number; unit: Caregivers
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 12
Caregivers | 12

4. Primary Outcome: Cultural Humility
Description: Caregivers will complete the Multicultural Therapy Competency Inventory- Client Version (MTCI-CV), adapted to assess perceptions of the Sleep Well! therapist's/program's cultural humility (e.g. "When we discussed my child's sleep, the Sleep Well! therapist seemed to have some understanding about my/my family's culture and background" and "When we discussed my child's sleep, the Sleep Well! therapist appreciated my expertise on my own life.") Average proportion of caregivers agreeing/strongly agreeing with statements on measure is reported.
Time Frame: 3 months
Population: The treatment evaluation form was administered at post-intervention only and was added to the protocol after feedback from family partners during the trial. Thus, data were not available for the 3 participants who did not complete the post-intervention assessment and the 2 participants that completed the intervention post-assessment before this measure was added.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 10
Participants
  Agree/strongly agree | 9
  Neutral | 1
  Disagree/strongly disagree | 0

5. Secondary Outcome: Sleep Patterns and Problems: Sleep Problem
Description: Caregivers will complete the Brief Child Sleep Questionnaire (BCSQ) to report on child sleep habits and the severity of any caregiver-perceived sleep problems at pretreatment and posttreatment. The BCSQ is appropriate for children ages 1.5-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child sleep.
Time Frame: Baseline (pre-intervention) and 3 months (post-intervention).
Population: Analysis was for those with both pre- and post-intervention data (N = 12)
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 12
Participants
  Reduction from sleep problem at pre to no sleep problem at post | 8
  Sleep problem at both pre and post | 4
Statistical Analysis 1: Comparison: Behavioral Sleep Intervention; Test type: Other; p = .008, McNemar — A priori statistical significance threshold = p<.05

6. Secondary Outcome: Sleep Patterns and Problems: Sleep Onset Latency
Description: Caregivers will complete the BCSQ to report on child sleep habits and the severity of any caregiver-perceived sleep problems at pretreatment and posttreatment. The BCSQ is appropriate for children ages 1.5-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep. When completing the BCSQ, caregivers are prompted to think about their child's sleep on a "typical night" over the past week (7 nights). Sleep onset latency is assessed by asking caregivers to report in minutes how long it typically takes their child to fall asleep.
Time Frame: 3 months
Population: Analysis was for those with both pre- and post-intervention data (N = 12)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 12
minutes
  Pre-intervention | 69.00 (50.41)
  Post-intervention | 25.83 (10.62)
Statistical Analysis 1: Comparison: Behavioral Sleep Intervention; Test type: Superiority; p = .014, t-test, 2 sided — A priori statistical significance threshold = p<.05

7. Secondary Outcome: Sleep Patterns and Problems: Night Awakening Duration
Description: Caregivers will complete the BCSQ to report on child sleep habits and the severity of any caregiver-perceived sleep problems at pretreatment and posttreatment. The BCSQ is appropriate for children ages 1.5-5 years and has shown good reliability and moderate correspondence with actigraphic recordings of child-sleep.
Time Frame: 3 months
Population: Analysis was for those with both pre- and post-intervention data, and with a corrected version of the BCSQ that included the duration of night awakenings question (N =7)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 7
minutes
  Pre-intervention | 131.25 (121.55)
  Post-intervention | 27.50 (58.56)
Statistical Analysis 1: Comparison: Behavioral Sleep Intervention; Test type: Superiority; p = .013, t-test, 2 sided — A priori statistical significance threshold = p<.05

8. Secondary Outcome: Sleep Patterns and Problems: Nighttime Sleep Duration
Description: as for outcome 7
Time Frame: 3 months
Population: Analysis was for those with both pre- and post-intervention data (N = 12)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 12
hours
  Pre-intervention | 6.63 (1.99)
  Post-intervention | 9.21 (1.21)
Statistical Analysis 1: Comparison: Behavioral Sleep Intervention; Test type: Superiority; p = .001, t-test, 2 sided — A priori statistical significance threshold = p<.05

9. Secondary Outcome: Sleep Patterns and Problems: 24-hour Sleep Duration
Description: as for outcome 7
Time Frame: 3 months
Population: Analysis was for those with both pre- and post-intervention data (N = 12)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Behavioral Sleep Intervention
Number analyzed (Participants) | 12
hours
  Pre-intervention | 8.71 (3.28)
  Post-intervention | 9.98 (1.03)
Statistical Analysis 1: Comparison: Behavioral Sleep Intervention; Test type: Superiority; p = .209, t-test, 2 sided — A priori statistical significance threshold = p<.05

ADVERSE EVENTS:
Time Frame: Through study completion; approximately 3 months
Arm/Group | Behavioral Sleep Intervention
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04046341/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT04046341/ICF_000.pdf